CLINICAL TRIAL: NCT06511024
Title: CASCADE: Profiling the Inflammatory Cascade of COVID-19
Brief Title: Profiling the Inflammatory Cascade of COVID-19
Acronym: CASCADE
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC20054
Record Dates: First submitted 2020-04-16; First posted 2024-07-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and other clinically available samples (e.g. BAL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: * Patients in the community
  * Patients at hospital admission
  * Rapidly deteriorating patients
  * Ventilated, critically ill patients With confirmed COVID-19 infection
  Interventions: Other: Blood sample
- Control: No clinical suspicion of COVID-19 infection
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Serial blood sampling to monitor immune cells in patient with COVID 19 infection and compare with control group who have no evidence of COVID-19 infection

SUMMARY:
COVID-19 is a new and poorly understood virus. It is imperative that the scientific community develops an understanding of the viral mechanisms and human immunological response in order to develop effective therapies and assess their efficacy.

This research study is being initiated in response to the ongoing COVID-19 pandemic and will provide much needed insight into the temporal immune response which can lead to rapid respiratory failure in infected patients.

DETAILED DESCRIPTION:
The immuno-inflammatory cascade is essential to define in COVID-19 patients to develop an intervention strategy to abrogate respiratory failure. For this study, four groups of patients have been identified to inform disease characterisation:

* Patients in the community
* Patients at hospital admission
* Rapidly deteriorating patients
* Ventilated, critically ill patients There is an urgent need to elucidate the dynamic peripheral blood signature including neutrophil, monocyte, lymphocyte and soluble mediators. Indeed recent data suggest that activation and subsequent exhaustion of cytotoxic T cells and emergence of GM-CSF+ CD4+ T cells and inflammatory monocytes and macrophages (in blood and BAL(1,2,3)) are associated with severe pathology in COVID-19 patients, however the fine kinetics of changes in these populations relative to disease progression are unknown.

In this study, samples will be obtained from NHS Lothian patients (in both primary care and hospital settings) who have tested positive for COVID-19 infection. Once consented, blood samples and (where possible) surplus clinical samples will be obtained from participants at defined time-points through the duration of their disease. Participants who rapidly deteriorate during their hospital admission will provide smaller, more frequent blood samples to permit profiling of the immunological/inflammatory response during deterioration.

Patients without COVID-19 but of comparable age and comorbid status will act as controls.

In-house assays will be used to measure and phenotype circulating immune cells, their activation status and cytokine production (focusing primarily on polymorphonuclear leukocytes, mononuclear phagocytes and lymphocytes) from peripheral blood samples obtained from participants at different stages of COVID-19 disease.

Blood and other clinical samples (including but not limited to Bronchoalveolar Lavage (BAL), bronchoabsorption) will undergo laboratory analysis, including but not limited to; whole blood cytokine release assays, inflammatory biomarkers and cell numbers, measurement of cytokines, flow cytometric cell analysis and staining of cells for markers.

Results will inform the identification of optimized biomarkers, timing of interventions and lead prioritisation of pharmaceutical assets for experimental medicine studies or assays for use in high throughput automated screens of compound libraries to modulate observed phenotypes and profile the inflammatory pathway. It will build from and complement emerging data from other national or international studies e.g. ISARIC 4C but will be distinct since it informs a specific translational study platform which requires greater depth of phenotyping and more precise kinetic analysis to inform design of early clinical studies of repurposed immunomodulating therapeutics. It is intended this will accelerate the linking of basic mechanistic information with drug targets for development and assessment of COVID-19 therapies. Research materials and results will be also be used to develop novel diagnostics and prognostic approaches that can help identify high risk patients who need higher level of monitoring or care and more fully define susceptibility and risk.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Aged over 16 years
* Provision of consent (either from the patient or by a personal legal representative)

COVID-19 Cohort only:

* Confirmed COVID-19 infection

Control Cohort only:

* No clinical suspicion of COVID-19

Exclusion Criteria:

All participants:

* Deemed unsuitable for participation by attending clinician

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort 1 COVID-19 Patients with confirmed COVID-19 infection (n=200) Cohort 2 Control Patients who have not tested positive for COVID-19 infection (n=20)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Determine levels of cytokines and chemokines to elucidate the temporal inflammatory cascade in COVID-19 | Up to 20 days
  We will determine levels of select cytokines and chemokines in plasma and serum samples from patients and control subjects.

SECONDARY OUTCOMES:
Identification, quantification and phenotyping of inflammatory cells and biomarkers. | Up to 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided